CLINICAL TRIAL: NCT03291054
Title: A Phase II Study of Epacadostat and Pembrolizumab in Patients With Imatinib Refractory Advanced Gastrointestinal Stromal Tumors
Brief Title: Epacadostat and Pembrolizumab in Patients With GIST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study ended prematurely at the request of the funding sponsor.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR1581
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumors; GIST; Pembrolizumab; Epacadostat; Columbia
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — pembrolizumab; spartalizumab; epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epacadostat and pembrolizumab (Experimental): Subjects will receive epacadostat and pembrolizumab
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat

INTERVENTIONS:
Drug: Pembrolizumab — Subjects will receive pembrolizumab 200 mg (flat dose) IV every 3 weeks on day 1 of a 21 day cycle.
  Other Names: Keytruda; Anti-PD-1 antibody
Drug: Epacadostat — Epacadostat will be dosed at 100 mg PO twice a day (BID) daily. Doses should be taken twice daily, in the morning and evening, approximately 12 hours apart, without regard to food.Doses will be self-administered, except on Cycle 2 Day 1, when the morning dose will be given at the study site clinic. Subjects will be required to keep a pill diary that will be provided to them.
  Other Names: INCB024360; IDO inhibitor

SUMMARY:
Primary objective is to assess the efficacy of combined Indoleamine 2,3-dioxygenase (IDO) and PD-1 inhibition in a single arm phase II trial of epacadostat and pembrolizumab in patients with advanced imatinib-refractory GIST, using a primary endpoint of overall response rate.

Secondary objectives are to evaluate the progression free survival (PFS), the overall survival (OS), the response rate and to evaluate the safety and tolerability of combined epacadostat and pembrolizumab treatment.

The investigator hypothesizes that treatment with epacadostat and pembrolizumab will increase the response rate compared to what has been historically achieved with salvage tyrosine kinase inhibitors.

DETAILED DESCRIPTION:
While targeted therapy with imatinib has significantly improved survival for patients with inoperable and metastatic gastrointestinal stromal tumors (GIST), the majority will eventually progress after a median of 20-26 months. Standard second-line treatment with sunitinib has a response rate of 7%, and third-line treatment with regorafenib has a response rate of only 5%. More effective treatments for imatinib-refractory GIST are needed.

This study aims to assess the efficacy of combined IDO and PD-1 inhibition with epacadostat (IDO inhibitor) and pembrolizumab (anti-PD-1 antibody) in patients with imatinib-refractory GIST.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of GIST.
* Unresectable or metastatic GIST
* Allowable prior therapies:

  1. Subjects must have had clinical or radiographic progression on imatinib. Those who were taken off of imatinib for intolerance must have progressed on at least one other tyrosine kinase inhibitor (TKI).
  2. Subjects must have received ≥ 1 prior systemic therapy (including imatinib). A maximum of 4 prior therapies for metastatic disease are allowed.
* Male or female subjects, age 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Life expectance of ≥ 3 months.
* Laboratory and medical history parameters within the following Protocol-defined range.

All screening laboratory tests should be performed within 28 days of treatment initiation and must be independent of hematopoietic growth factor support.

* Absolute neutrophil count ≥ 1.5 x 109/L.
* Platelets ≥ 100 x 109/L.
* Hemoglobin ≥ 9 g/dL (transfusion is acceptable to meet this criteria)
* Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN) OR calculated creatinine clearance ≥ 50 mL/min for subjects with creatinine levels > 1.5 x institutional ULN.
* Aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase ≤ 2.5 x ULN, or ≤ 5 x ULN in subjects with liver metastases.
* Total bilirubin ≤ 1.5 x ULN

  o Note: patients with hyperbilirubinemia clinically consistent with an inherited disorder of bilirubin metabolism (eg, Gilbert syndrome) will be eligible at the discretion of the principal investigator.
* International normalized ratio (INR) or prothrombin time (PT) < 1.5x ULN unless subject is receiving anticoagulation therapy as long as PT or INR is within therapeutic range of intended use of anticoagulant.
* Activated partial thromboplastin time (aPTT) < 1.5 x ULN unless subject is receiving anticoagulant therapy, as long as PTT is within therapeutic range of intended use of anticoagulants.

  * Presence of baseline measureable disease by RECIST v1.1 for solid tumors, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan, MRI, or calipers by clinical exam. (See Section 15.4 for the evaluation of measurable disease).
  * The effects of pembrolizumab and epacadostat on the developing human fetus are unknown, and thus female subjects of childbearing potential (defined as women who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy, and are not postmenopausal (defined as ≥ 12 months of amenorrhea)) must have a negative pregnancy test at screening and must agree to use adequate contraception (complete abstinence, or two methods of birth control (Appendix B)) prior to study entry and until at least 4 months after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * Fertile men must also agree to use adequate contraception (2 barrier methods or abstinence) during the study and for up to 4 months after the last dose of study drug.
  * All subjects must agree to pre- and on-treatment tumor biopsies. Subjects in whom biopsy is technically not feasible or in whom would result in unacceptable risk, in the opinion of the investigator, may be exempted from the biopsy requirement with discussion with the principal investigator. Use of outside archived tumor tissue for a baseline biopsy is not permitted.
  * Willingness and ability to provide written informed consent prior to any study-related procedures and to comply with all study requirements.

Exclusion Criteria:

* Treatment with chemotherapy (not including Tyrosine Kinase Inhibitors) or radiotherapy within 4 weeks (6 weeks from nitrosoureas or mitomycin C), or treatment with monoclonal antibody therapy within 4 weeks prior to start of study treatment. Note: No minimum washout period is required for tyrosine kinase inhibitor therapy (eg, imatinib or sunitinib).
* Patients must have recovered from adverse events (greater than grade 1) due to prior anticancer therapy, except for stable chronic toxicities such as alopecia.
* Participation in any other clinical study with investigational drug received within 28 days or 5 half lives (whichever is longer) before first dose.
* Subjects who have received prior anti-PD-1 or anti-PD-L1 antibody, or an IDO inhibitor.
* Subjects who have received experimental vaccines or other immune therapies should be discussed with the principal investigator to confirm eligibility.
* Any prior ≥ Grade 3 immune-related adverse event (irAE) while receiving immunotherapy, or any unresolved irAE > grade 1.
* Subjects receiving immunologically based treatment for any reason, including chronic steroids or prednisone (at dose >10 mg/day of prednisone) within 14 day prior to first study treatment. Inhaled or topical steroids or systemic steroids (at dose ≤10 mg/day of prednisone) is permitted.
* Subjects with any active or inactive autoimmune process (eg, rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease) or who are receiving systemic therapy for an autoimmune disease. Exceptions include vitiligo, hypothyroidism controlled on hormone replacement, type I diabetes, Grave's disease, adrenal insufficiency on stable replacement doses of steroids (prednisone ≤10 mg/day or equivalent), or with principal investigator approval.
* No prior organ allograft or allogenic bone marrow transplantation.
* History of (noninfectious) pneumonitis that require steroids or current pneumonitis.
* A diagnosis of another active malignancy with the following exceptions: basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, isolated elevation of prostate-specific antigen, indolent secondary malignancies not requiring active therapy, or with the approval of the principal investigator. Subjects with a completely treated prior malignancy and no evidence of disease for ≥ 2 years are eligible.
* Subjects with known active hepatitis B (HBV) or hepatitis C (HCV) infection as defined by the following (Hepatitis screening studies are required:

  * Positive test for hepatitis B surface antigen
  * Positive test for hepatitis C antibody and/ or hepatitis C quantitative viral load (Note: Subjects with a positive hepatitis C antibody and negative quantitative hepatitis C polymerase chain reaction (PCR) viral load are eligible)
* Subjects with a known history of HIV, including patients with controlled disease on antiretroviral therapy. HIV testing is not required as part of screening for this study.
* Subjects receiving monoamine oxidase (MAO) inhibitors within 21 days of study enrollment (epacadostat increases serotonin levels, theoretically increasing the risk of serotonin syndrome, although this has not been reported in any ongoing clinical studies to date).
* Any history of serotonin syndrome (SS) after receiving 1 or more serotonergic drugs.
* Current pregnancy or breast feeding. Pregnant women are excluded from this study because the teratogenicity of epacadostat and pembrolizumab are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab and/or epacadostat, breastfeeding should be discontinued in all female subjects.
* Receipt of live attenuated vaccines (including, but not limited to: intranasal influenza vaccine (FluMist), measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine) within 30 days before the first dose of study treatment.
* Concurrent use of any medication that is an inhibitor of UGT1A9 during the screening or treatment period.
* Major surgical procedure or significant traumatic injury within 14 days of initiating study drug or anticipation of the need for major surgery during the study.
* Inability to swallow capsules, or refractory nausea and vomiting, malabsorption, an external biliary shunt, or significant bowel resection that would preclude adequate absorption.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, active liver disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, or interfere with the subject's participation for the full duration of the study.
* Known allergy or reaction to any component of either study drug formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Carvajal, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - U-M Comprehensive Cancer Center, Ann Arbor, Michigan
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Epacadostat and Pembrolizumab
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Data was not analyzed or disclosed in an effort to protect subject confidentiality (n=1).
Arm/Group | Epacadostat and Pembrolizumab
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The primary endpoint is the overall response rate as defined as the best response using RECIST v1.1 criteria. A standard way to measure how well a cancer patient responds to treatment. It is based on whether tumors shrink, stay the same, or get bigger. To use RECIST, there must be at least one tumor that can be measured on x-rays, CT scans, or MRI scans. The types of response a patient can have are a complete response (CR), a partial response (PR), progressive disease (PD), and stable disease (SD). Also called Response Evaluation Criteria In Solid Tumors.
Time Frame: within the first 24 weeks of the start of study therapy
Population: Data was not analyzed or disclosed in an effort to protect subject confidentiality (n=1).
Arm/Group | Epacadostat and Pembrolizumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Description: The length of time from the start of treatment that patients diagnosed with the disease are still alive.
Time Frame: time from registration up to 2 years
Population: Data was not analyzed or disclosed in an effort to protect subject confidentiality (n=1).
Arm/Group | Epacadostat and Pembrolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Days 1, 8, and 15 of cycle 1 and day 1 of all subsequent cycles. Data was not analyzed or disclosed in an effort to protect subject confidentiality (n=1).
Arm/Group | Epacadostat and Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the complete nor any part of the results of the study carried out under this protocol, nor any of the information provided by the sponsor for the purposes of performing the study, will be published or passed on to any third party without the consent of the study sponsor. Any investigator involved with this study is obligated to provide the sponsor with complete test results and all data derived from the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT03291054/Prot_SAP_000.pdf